CLINICAL TRIAL: NCT06649786
Title: Comparison of the Efficacy and Safety of Endoscopic Hemorrhoids Ligation: a Single-center Randomized Controlled Clinical Trial
Brief Title: Comparison of the Clinical Efficacy and Safety of Endoscopic Superior Rectal Mucosal Ligation and Hemorrhoids Ligation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QYFYEC2024-137
Record Dates: First submitted 2024-10-17; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-10

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic superior rectal mucosal ligation group (Experimental): The patient is treated with endoscopic superior rectal mucosal ligation
  Interventions: Procedure: Endoscopic superior rectal mucosal ligation
- Endoscopic hemorrhoid ligation group (Active Comparator): The patient is treated with endoscopic hemorrhoids ligation
  Interventions: Procedure: Endoscopic hemorrhoid ligation

INTERVENTIONS:
Procedure: Endoscopic superior rectal mucosal ligation — The patient takes the left side decubitus position, the endoscope is connected with 6 serial ligators, the cup of the sleeve is pointed at the upper edge of the straight anal line and the rectal mucosa is continuously aspirated under negative pressure. The mucosa enters the sleeve and sees a full-screen red sign. The sensing loop is successfully triggered, indicating that the loop is complete.
  Arms: Endoscopic superior rectal mucosal ligation group
Procedure: Endoscopic hemorrhoid ligation — The patient takes the left side decubitus position,the endoscope is connected with 6 serial ligators,the cup the sleeve is aligned with the base of the hemorrhoid (above the dentate line) for continuous negative pressure suction.The hemorrhoid enters the sleeve and sees a full-screen red sign. Turn the handle of the sleeve clockwise and feel that the loop is successfully triggered, the ligature is completed.
  Arms: Endoscopic hemorrhoid ligation group

SUMMARY:
Endoscopic superior rectal mucosal ligation and hemorrhoids ligation are two types of endoscopic ligation, The aim of this study is to compare the clinical efficacy and safety of these two approaches.If you accept this study,you need to provide case information before the operation, complete the endoscopic treatment according to the routine colonoscopy procedure, and follow-up survey after the operation.

ELIGIBILITY:
Inclusion Criteria:

1. According to the Goligher classification in the Chinese guidelines for the diagnosis and treatment of hemorrhoids (2020) , patients who are diagnosed with grade II-III internal hemorrhoids .
2. Patients who voluntarily participate and sign the informed consent form.

Exclusion Criteria:

1. patients who had severe heart, liver, and kidney disease.
2. patients who had severe immune deficiency.
3. patient's general condition is too poor to tolerate endoscopic therapy.
4. patients had a history of pelvic chemoradiotherapy.
5. patients had severe infection or inflammatory lesion in the rectum or anal canal,or the rectum or anal canal had undergone surgery.
6. patient is a pregnant woman.
7. patients who disagree with endoscopic treatment and are concerned about the possible risks refused to sign the informed consent form.
8. the follow-up time is insufficient and the clinical data were incomplete.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 96 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
complication | 7 days after operation
  Postoperative complications, such as dysuria, thrombotic external hemorrhoids, perianal abscess,and so on.
clinical efficacy | 1 month after operation
  Complete disappearance of postoperative symptoms is regarded as a cure, postoperative symptoms relief is regarded as partial cure, and symptoms as same as before are considered ineffective.

IPD SHARING:
Plan to Share IPD: Yes
The statistical results of the clinical data collected in the experiment (baseline characteristics, preoperative disease-related data, postoperative disease-relate）will be shared.